CLINICAL TRIAL: NCT01667874
Title: Use of Collatamp G Antibiotic Impregnated Sponges in the Treatment of Peri-prosthetic Total Joint Infections
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulty in recruiting patients for the study
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Richard McCalden, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 102635
Record Dates: First submitted 2012-08-15; First posted 2012-08-17 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Infection
Keywords: Randomized controlled trial; early joint infection; gentamicin impregnated sponges
MeSH Terms: conditions — Infections | interventions — Gentamicins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Collatamp sponge (No Intervention): Joint infection treated without the use of the Collatamp G sponge.
- Collatamp G sponge (Experimental): Use of Collatamp G Gentamicin impregnated sponge for the treatment of early total joint infections
  Interventions: Drug: Collatamp G sponge

INTERVENTIONS:
Drug: Collatamp G sponge — Collatamp G is an antibiotic impregnated sponge
  Other Names: Gentamicin Sulphate 2.0 mg/cm2
  Arms: Collatamp G sponge

SUMMARY:
The purpose of this study is to determine if Collatamp, a small flat sponge soaked with antibiotics will help to improve the success rate of the treatment of acute joint infections after a joint replacement surgery. Our hypothesis is that those patients receiving the Collatamp sponges will have an improved success with respect to the eradication of infection at one year following treatment.

DETAILED DESCRIPTION:
While total hip and knee replacement surgery remains a highly successful treatment for arthritis of the hip and knee, infection following a joint replacement still remains an issue, occurring in approximately 1-2% of joint replacement patients. Treatment of infection remains very difficult with the successful elimination of the infection being quite variable, ranging from as low as 10% to approximately 85-90%, following a two stage revision. A two stage revision involves removing the joint replacement implant and replacing it with a cement spacer until the surgeon is comfortable that the infection has been eliminated. In the second part of a two stage revision the cement spacer is removed and a new joint replacement implant is inserted in the joint space. In particular, the treatment of an acute infection, that is, infection occurring in the early postoperative period or in a patient with less than two weeks duration of symptoms, is particularly problematic. As a first line of treatment, surgeons often perform an irrigation (washing out a wound with a stream of water) and debridement (the surgical removal of contaminated tissue) surrounding the joint in the hopes of preserving the joint replacement, although the success rate is highly variable. Most treatment routines involve irrigation of the joint with copious (large) amounts of fluid, removal of infected soft tissue, replacement of any removable parts (example plastic liners or femoral heads) and then intravenous antibiotics for a prolonged period of time (6-8 weeks). It is thought that part of the reason for failure with this form of treatment is the inability to adequately provide local antibiotics to the joint environment while the joint replacement components are in place. In particular, the formation of a bacterial slime by the infecting organism, which can attach itself to the metallic components, is thought to be a major hindrance to removing infection. In theory, the ability to infuse local antibiotics to the joint could prove advantageous to the treatment of joint replacement infections.

Collatamp® is a like a small flat sponge soaked with antibiotics that delivers a consistent dose of fast-release antibiotics called Gentamicin Sulphate (2.0 mg/cm2). The antibiotic is concentrated locally in the tissue around the joint replacement. The sponge is reabsorbed by the body and therefore does not need to be surgically removed. Collatamp® sponges have been utilized in the clinical setting for over 20 yrs. This material has been used in treatment of other orthopaedic, general surgery, and cardiac infections, but has not been studied in the setting of infected total joint replacements. The purpose of this study is to examine the use of CollatampTM sponges as an addition to the treatment of acute joint infections after a total joint replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an acute total joint infection

Exclusion Criteria:

* History of alcoholism
* Unable to return for follow-up
* Refuses to participate in the study
* Does not speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
Eradication of infection | One year
  Success will be defined as those patients whose implant is still in place at one year and demonstrate no clinical signs or symptoms of infection. Eradication of infection will be defined as those patients whose inflammatory markers (ESR and CRP)have returned to normal values following one year treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Richard McCalden, MD, MPhil(Edin), F.R.C.S.(C), Principal Investigator — London Health Sciences Centre - University Hospital
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stemberger A, Grimm H, Bader F, Rahn HD, Ascherl R. Local treatment of bone and soft tissue infections with the collagen-gentamicin sponge. Eur J Surg Suppl. 1997;(578):17-26. No abstract available. PMID 9167145